CLINICAL TRIAL: NCT05725590
Title: A Multicenter Randomized Controlled Study of External Pancreatic Duct Stents in Pancreaticoduodenectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Ningbo No. 1 Hospital (Other); Huizhou Municipal Central Hospital (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); The Third Affiliated Hospital of Wenzhou Medical University (Other); Linping First People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-0976
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Pancreatic Fistula
Keywords: Clinically relevant postoperative pancreatic fistula; External pancreatic duct stent; Pancreaticoduodenectomy
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- external pancreatic duct stent (Experimental)
  Interventions: Procedure: External pancreatic duct stent
- internal pancreatic duct stent (Experimental)
  Interventions: Procedure: Internal pancreatic duct stent

INTERVENTIONS:
Procedure: External pancreatic duct stent — All pancreaticoduodenectomies were performed by the same surgical team at our pancreatic center throughout the study period. According to the preoperative laboratory results, medical imaging data, and intraoperative conditions, the laparoscopic or open pancreaticoduodenectomy, or pylorus-preserving pancreaticoduodenectomy was performed at the discretion of the individual surgeon. The child's technique was implemented to achieve digestive tract reconstruction, and all patients underwent a duct-to-mucosa pancreaticojejunostomy. The external pancreatic duct stent left the other end exteriorized through the proximal jejunum via a small enterotomy that was fixed in the abdominal wall.
  Arms: external pancreatic duct stent
Procedure: Internal pancreatic duct stent — All pancreaticoduodenectomies were performed by the same surgical team at our pancreatic center throughout the study period. According to the preoperative laboratory results, medical imaging data, and intraoperative conditions, the laparoscopic or open pancreaticoduodenectomy, or pylorus-preserving pancreaticoduodenectomy was performed at the discretion of the individual surgeon. The child's technique was implemented to achieve digestive tract reconstruction, and all patients underwent a duct-to-mucosa pancreaticojejunostomy. The internal pancreatic duct stent, a silicone catheter with multiple side pores, was inserted into the main pancreatic duct and the other end was placed in the jejunum cavity.
  Arms: internal pancreatic duct stent

SUMMARY:
The prognostic value of external vs internal pancreatic duct stents after pancreaticoduodenectomy remains controversial. This study aimed to evaluate the benefits of external and internal stents using the Updated Alternative Fistula Risk Score in both high-risk and low-risk patients with regard to the incidence of clinically relevant postoperative pancreatic fistula.

DETAILED DESCRIPTION:
Pancreatic cancer, with its associated poor prognosis, is one of the most insidious and lethal cancers globally. Indeed, pancreatic cancer has been listed as the fourth leading cause of cancer-related deaths in developed countries, and it may replace colorectal cancer as the second-leading cause of cancer-related deaths by 2030. Pancreaticoduodenectomy is the standard treatment for periampullary carcinoma, especially pancreatic head tumors. However, the incidence of postoperative complications, especially postoperative pancreatic fistula, remains as high as 25%-50%, which limits the dissemination of pancreaticoduodenectomy.

An external pancreatic duct stent is one of the methods used to prevent pancreatic fistula. A large number of studies, including prospective randomized trials as well as meta-analyses, have shown that external pancreatic duct stents significantly decrease the rate of pancreatic fistula and shorten the length of hospital stay. Paradoxically, several studies have shown that external pancreatic duct stents have no effect and may even increase the incidence of postoperative pancreatic fistula. In a meta-analysis, Dong et al. observed that the use of an external pancreatic duct stent was associated with a significantly lower incidence of pancreatic fistula in patients at high risk for pancreatic fistula compared with an internal stent, but there was no definitive conclusion because of the low quality of the evidence.

In 2019, Mungroop et al. proposed the Updated Alternative Fistula Risk Score (ua-FRS) according to the International Study Group of Pancreatic Surgery (ISGPS), which quantitatively validated the risk of pancreatic fistula and assessed the benefits of pancreatic duct stents in patients at different levels of risk. Moreover, ISGPS redefined the classification criteria for pancreatic fistula (Grade A) as a biochemical leak, which had no significant clinical impact on the clinical prognosis. In addition, the position statement by ISGPS indicated that, due to the lack of high-quality evidence, the pancreatic duct stent was not routinely recommended during pancreaticoenteric anastomosis, but external stenting can be considered in high-risk glands. Therefore, it is necessary to systematically re-investigate the safety and effectiveness of external pancreatic duct stents for the prevention and treatment of clinically relevant postoperative pancreatic fistula (CR-POPF) in both high-risk and low-risk patients. This retrospective study was conducted to evaluate the differences between external and internal pancreatic stents using the ua-FRS scoring system, based on the hypothesis that the use of an external stent in high-risk patients could decrease the rates of CR-POPF compared with an internal stent after pancreaticoduodenectomy.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatoduodenectomy with pancreaticojejunal mucosa anastomosis was performed;

  * The patient has no combined organic diseases in the heart, lungs, or kidneys;

    * No history of chemotherapy, radiotherapy, upper abdominal surgery, or combined with other tumors; ④ The risk score of the pancreatic fistula of the patient according to the definition of the updated Alternative Fistula Risk Score (ua-FRS). Patients with a ua-FRS score higher than 5% were included in this study.

Exclusion Criteria:

* Previous history of other tumors or upper abdominal surgery; ② Multiple lesions and distant metastasis;

  * Patients with organic diseases of important organs such as the heart, lung, and kidney, who cannot tolerate surgery, or patients who are more than 75 years old or less than 18 years old; ④ Other measures were performed to prevent pancreatic fistula, such as fibrin glue sealing, which may affect the accuracy of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
The incidence of CR-POPF | 1 month after the surgery completion
  The primary endpoint of this retrospective study was the incidence of CR-POPF, which was graded according to the definition set forth by ISGPS in 2016.

SECONDARY OUTCOMES:
The incidence of other complications | 1 month after the surgery completion
  The secondary endpoints of this retrospective study included the incidence of delayed gastric emptying (DGE), postoperative pancreatic hemorrhage (PPH), bile leakage, infection and mortality, which were graded according to the Clavien-Dindo Classification.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Yan, Doctor, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China; Yuancong Jiang, Doctor, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available from the author on reasonable request.